CLINICAL TRIAL: NCT05883293
Title: Clinical Study of Allogeneic Fat Decellularized Active Protein in the Treatment of Pulmonary Fibrosis
Acronym: CEFFE-PF
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEFFE-PF-2023
Record Dates: First submitted 2023-04-18; First posted 2023-05-31 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Fibrosis
Keywords: Cell Free Fat Extract ，CEFFE; Pulmonary Fibrosis; nebulized inhalation
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Case Inclusion Criteria:
  1. Patients who sign the informed consent form.
  2. Age 30~80 years old, gender is not limited.
  3. Patients with pulmonary fibrosis who have obvious pulmonary fibrosis symptoms, signs, and HRCT abnormalities, and are diagnosed as pulmonary fibrosis patients specified in this protocol, and have poor effect of existing treatment regimens or do not accept existing treatment regimens
  Clinical basis for diagnosis of pulmonary fibrosis:
  1. Abnormal pulmonary function, including restrictive ventilatory dysfunction and gas exchange disorder;
  2. Typical fibrotic manifestations on HRCT: such as interstitial changes, grid-like changes or honeycomb lungs;
  Interventions: Drug: Cell Free Fat Extract(CEFFE)

INTERVENTIONS:
Drug: Cell Free Fat Extract(CEFFE) — The subjects inhaled 2ml of CEFFE each time in a nebulized inhalation method, inhaling every 3 days, for a total of 7 inhalations

SUMMARY:
The purpose of this clinical trial is to investigate the efficacy and safety of allogeneic adiphatic cyclic active protein in the treatment of pulmonary fibrosis.

The main questions it aims to answer are:

1. Efficacy of allogeneic adiposeactive protein in the treatment of pulmonary fibrosis
2. Safety of allogeneic fat respiration active protein in the treatment of pulmonary fibrosis.

A total of 7 participants will be enrolled. Participants will be asked that they will receive 2ml of each nebulized inhalation Cell Free Fat Extract (CEFFE), inhaled every 3 days, for a total of 7 nebulized inhalation treatments.

The clinical trial was designed using a single-center, self-controlled trial with no control group and no blinding.

DETAILED DESCRIPTION:
1. Research purpose:

   Main Objective: To study the efficacy and safety of allogeneic adiphacyclic active protein in the treatment of pulmonary fibrosis, the main observation and evaluation indicators included: clinical efficacy, clinical adverse events and abnormal laboratory tests.

   The basis of the question:

   Animal experiments have found that fat decellularization active protein has a certain improvement effect in bleomycin-induced mouse pulmonary fibrosis model. At present, domestic clinical studies have found that fat acellular active protein is safe for the treatment of human diseases and has no obvious side effects. Therefore, in this study, the allogeneic adipo-decellularized active protein was treated with aerosol inhalation in the treatment of pulmonary fibrosis to observe its efficacy and safety.
2. Research Design:

   Overall design: Single-center, self-controlled experimental design was adopted, no control group was set up, and no blinding method was adopted.

   Number of planned cases: 7.

   Indications: Pulmonary fibrosis.
3. Clinical trails process:

   3.1 Sign the informed consent form and collect relevant clinical data; For patients with a definitive diagnosis of pulmonary fibrosis

   3.2 Allogeneic Cell Free Fat Extract (CEFFE) treatment process:

   3.2.1 Preparation of CEFFE of allogeneic origin

   Healthy donors who underwent liposuction at the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine signed a written informed consent form. Under local anesthesia, a healthy donor injects swollen fluid into the abdomen, and operates with a 20mL syringe or a mechanical negative pressure machine (laser, ultrasound, microwave and other assisted liposuction methods cannot be added), and the group is determined according to the sequence of enrollment from low to high, and the fat is extracted according to the required dose, and the amount of liposuction in a single session should be 150ml -200ml. The collected adipose tissue is rinsed with normal saline, left to stand, and centrifuge at 1200g for 3 minutes. At the end of centrifugation, remove excess water from the bottom end, collect them separately in sterile 50mL syringes for storage and transfer. Adipose tissue active factors are prepared in the laboratory and cryopreserved. Two 10mL syringes connected by tee tubes, mechanically emulsified 60 times, collected into 50mL centrifuge tubes, centrifuged at 2000g for 5min. After centrifugation, the bottom clear liquid layer was collected, filtered through a 0.22um filter, and the fat decellularized active protein was obtained, which was frozen in a -20°C freezer.

   3.2.2 Health Donor Selection Criteria:

   3.2.2.1 Age 18-45, male or female

   3.2.2.2 Liposuction at the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine

   3.2.2.3 Sign the informed consent form for biological sample donation

   3.2.3 Exclusion Criteria:

   3.2.3.1 Patients with hepatitis B, hepatitis C, HIV, syphilis, cytomegalovirus, herpesvirus and other infections

   3.2.3.2 Patients with severe hypertension, diabetes, heart disease and other chronic diseases

   3.2.3.3 Patients with tumors or previous history of tumors

   3.3 After negative percutaneous test, allogeneic CEFFE is inhaled by nebulization; 0.2ml CEFFE was injected intradermally 1 cm above the palmar stria on the palmar side of the right forearm, and 0.2ml of normal saline was injected intradermally 1 cm above the palmar stria on the palmar side of the left forearm as a control. Interpretation of skin test results: local pichu bulge, and red halo hard lump, diameter > 1 cm is positive.

   Give a single dose of 2ml allogeneic CEFFE stock solution (protein concentration of 3mg/ml), administered by nebulization inhalation, 8 minutes between each atomization time, 3 days apart; A total of 7 doses were given.

   3.4 The clinical symptoms, chest CT, lung function and related adverse reactions were observed at 1 month, 3 months, 6 months and 12 months after allogeneic fat decellularization active protein treatment.
4. Evaluation Criteria:

   4.1 Efficacy criteria:

   4.1.1 Obvious effect means that the main symptoms and signs are significantly relieved, and the objective indicators are significantly improved.

   4.1.2 Effective means that the main symptoms and signs have improved, and the objective indicators have improved.

   4.1.3 Ineffective means that the main symptoms and signs have not changed, and the objective indicators have not changed significantly or worsened.

   4.2 Safety evaluation:

   Clinical adverse events and laboratory tests are definitely related to allogeneic CEFFE treatment, likely related to allogeneic CEFFE treatment, may be related to allogeneic CEFFE treatment, may not be related to allogeneic CEFFE treatment, and may not be related to allogeneic CEFFE treatment.

   4.3 Evaluation endpoints: Clinical efficacy, comprehensive efficacy and safety evaluation at 1, 3, 6 and 12 months after the end of treatment were the main evaluation endpoints.
5. Quality assurance of clinical trial data

   The quality control of this clinical trial is controlled and controlled by the Ninth People's Hospital affiliated to Shanghai Jiao Tong University School of Medicine, and the research work is carried out in accordance with GCP, SOP and quality control requirements. Develop a clinical research plan. GCP training for relevant researchers participating in the trial.

   5.1 Before the start of the trial, the plan should be submitted to the Ethics Committee of the Ninth People's Hospital affiliated to Shanghai Jiao Tong University School of Medicine for approval;

   5.2 in accordance with GCP guidelines, necessary steps should be taken during the design and implementation phases of the study to ensure that the data collected is accurate, consistent, complete and credible;

   5.3 The participating researchers will strictly follow China's GCP standards to conduct the trial, collect and record the contents of the case report form truthfully, carefully and in detail in accordance with the clinical trial standard operating procedures (SOP), and verify them to ensure the reliability of the data;

   5.4 The investigator fills in the information required by the protocol into the Case Report Form (CRF), and the supervisor verifies that it is complete and accurate, and instructs the staff of the research center to make necessary corrections and supplements;

   5.5 All kinds of instruments, equipment, reagents, standards, etc. used in various inspection items in clinical trials should have strict quality standards and ensure that they work under normal conditions;

   5.6 Send statistical issues in the test plan to statistical experts for review and check;

   5.7 During the trial, the investigator monitors the research process, informed consent, and the correctness and completeness of the data in the case report form (CRF).
6. Recording and preservation of research materials

   In accordance with the GCP principle, the investigator should keep all the detailed original files of the subjects, and record the relevant test process, medication, laboratory test data, safety data and efficacy evaluation in the case report form, and the recorded data should be complete, timely and clear. Case report forms, original documents, medical records, etc. should be clear, detailed and easily identifiable by personnel participating in this clinical trial.

   At a minimum, the principal investigator must sign the inclusion confirmation page and completion page of the case report form to confirm the accuracy and completeness of all data.

   The case report form and the original file can only be modified by the investigator. Any changes to the case report form and the original file must not erase the original data. The correct modification method is to draw a single line on the original data, and then write the modified data next to the original data, and sign the date and the initials of the person who modified it.

   Test data should be retained for 10 years after the end of the test. However, if required by current regulations or agreements with sponsors, these data should be kept for a longer period of time.
7. statistical treatment scheme

   7.1 filling in the case report form (CRF) The investigator should complete the filling of case report form in time, modify it according to the correct modification method, and the completed case report form shall be reviewed and signed by the main researchers

   7.2 statistical analysis method and statistical description

   7.2.1 Treatment of missing value of main efficacy index data: when some subjects lack a major efficacy data, the method of filling deficiency is determined from the statistical and professional perspective. If the case is missing, the data of the previous measurement shall be transferred.

   7.2.2 Case analysis of incomplete test: the reasons for exfoliation should be analyzed one by one.

   7.2.3 Descriptive statistics: mean, standard deviation, maximum value, minimum value, median, confidence interval, frequency (composition ratio), etc.

   7.3 Statistical expression

   7.3.1 The report mainly uses tables to show that the tables are self-evident, that is, they have table questions, table notes and examples.

   7.3.2 The results of repeated measurement data are expressed in tables and statistical charts are attached to increase readability.

   7.4 Statistical software SAS 9.1.3 and Das for clinical trial 3.0 software were used to analyze the software simultaneously, and the results were confirmed.
8. Modification and interim analysis in the course of the test

Once the research plan has been discussed by the research group and reviewed by the ethics committee, it is not allowed to change at will; before the modification is implemented, the researcher must report the content and reason of the modification to the ethics committee of clinical trial for approval, and then carry out the research according to the modified scheme.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign the informed consent form.
2. Age 30~80 years old, gender is not limited.
3. Patients with pulmonary fibrosis who have obvious pulmonary fibrosis symptoms, signs, and HRCT abnormalities, and are diagnosed as pulmonary fibrosis patients specified in this protocol, and have poor effect of existing treatment regimens or do not accept existing treatment regimens

Clinical basis for diagnosis of pulmonary fibrosis:

1. Abnormal pulmonary function, including restrictive ventilatory dysfunction and gas exchange disorder;
2. Typical fibrotic manifestations were found on HRCT, such as interstitial changes, grid-like changes or honeycomb lungs

Exclusion Criteria:

1. Patients suffering from any of the following diseases: active tuberculosis, lung abscess, aspiration pneumonia, lung tumor, pulmonary edema, atelectasis, pneumothorax, pleural effusion, pulmonary embolism, pulmonary eosinophilic infiltration, pulmonary vasculitis and immunosuppression or immunodeficiency (including: hepatitis B surface antigen, hepatitis C antibody, AIDS antibody, syphilis antibody test positive);
2. Patients with active infection within 4 weeks;
3. Patients with acute exacerbation of pulmonary fibrosis within 4 weeks or/and those who require high-flow oxygen (oxygen concentration greater than or equal to 40% or oxygen flow greater than or equal to 5L/min), non-invasive or invasive ventilator-assisted ventilation
4. Patients with a history of tumor or current tumors;
5. The patient has a severe life-threatening disease and is expected to survive less than 12 months;
6. The patient has leukopenia (neutrophil count< 1000/mm3);
7. Patients with severe renal impairment: creatinine clearance < 30ml/min/1.73m2 or serum creatinine >265μmol/L (>3mg/dL);
8. Patients with liver disease or severe liver function impairment: ALT, AST > 2 times the upper limit of normal value;
9. Those with central nervous system dysfunction, such as convulsions, impaired consciousness, history of epilepsy or seizures; Have a clear history of mental disorders, or a history of psychotropic substance abuse or drug abuse
10. Long-term use of glucocorticoids for treatment of more than 10 mg of prednisone or equivalent, immunosuppressants or antifibrotic drugs, such as penicillamine, colchicine, cyclosporine A, TNFα antagonists, imatinib, IFN-γ, azathioprine, cyclophosphamide;
11. Women who are pregnant, breastfeeding or do not use proper contraception;
12. Those who are allergic to known ingredients of drugs and who are known or suspected of being allergic to the active or inactive ingredients of the study drug;
13. Allergy to acetaminophen or history of hypersensitivity reactions;
14. Alcohol abuse (defined as drinking >2 units per day/1>4 units per week, drinking 1 unit equivalent to 360ml of beer or 45ml of spirits with 40% alcohol content or 150ml of wine) or drug abusers;
15. Any situation that the investigator believes may increase the risk of the patient or interfere with the clinical trial, and the patient is not suitable for entering the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Modified UK Medical Research Council Respiratory Questionnaire (mMRC) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  The change of mMRC at each time node
Borg grading scale | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  The change of Borg grading scale at each time node
SGRQ Quality of Life Questionnaire | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  The change of SGRQ at each time node

SECONDARY OUTCOMES:
Vital capacity (VC) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  The change of VC at each time node
Forced vital capacity (FVC) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  The change of FVC at each time node
Forced expiratory volume in the first second (FEV1) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  The change of FEV1 at each time node
The ratio of the measured carbon monoxide dispersion to the expected value (DLCO%) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  The change of DLCO at each time node
Adverse reactions | 1 month, 3 months, 6 months, 12 months after treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 at each time node
6-minute walk test | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  Change in walking distance in 6-minute walk test
Pressure of oxygen in blood gases | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  The change of pressure of oxygen in blood gases
Complete blood count(Safety and tolerability) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  Complete blood count
Alanine aminotransferase(Safety and tolerability) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  Alanine aminotransferase
aspartate aminotransferase(Safety and tolerability) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  aspartate aminotransferase
r-glutamyl transferase(Safety and tolerability) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  r-glutamyl transferase
alkaline phosphatase(Safety and tolerability) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  alkaline phosphatase
creatinine(Safety and tolerability) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  creatinine
urea nitrogen(Safety and tolerability) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  urea nitrogen
uric acid(Safety and tolerability) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  uric acid
electrocardiogram(Safety and tolerability) | baseline; 1 month, 3 months, 6 months, 12 months after treatment
  Presence or absence of ECG abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- The Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No